CLINICAL TRIAL: NCT03114059
Title: Retro- and Prospective Monocentric Study to Evaluate the Safety and Effectiveness of the CyPass Stent 5 Years After Implantation
Brief Title: 5 Years Long Term Results After Standalone CyPass-Implantation
Status: Completed | Type: Observational
Sponsor: Dietrich-Bonhoeffer-Klinikum (Industry)
Responsible Party: Sponsor
Other Study IDs: STI 06/16
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2018-08

CONDITIONS: Glaucoma
Keywords: Late Effects of Surgery
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- standalone CyPass implantation: patients who have undergone a standalone cypass implantation without cataract surgery more than 3 years ago
  Interventions: Diagnostic Test: Glaucoma diagnostics

INTERVENTIONS:
Diagnostic Test: Glaucoma diagnostics — Heidelberg Retinal Topography, Visual field, intraocular pressure, medication anamnesis, Retinal Nerve Fibre Layer Thickness, Pachymetry, Sonography, full ophthalmological examination

SUMMARY:
This study evaluates the results of all clinically relevant findings of glaucoma diagnostics 5 Years after stent-implantation concerning the safety and effectiveness of the cypass stent procedure. The comparison of Preoperative and long term postoperative results is the aim of this study to evaluate this young procedure of Glaucoma surgery

DETAILED DESCRIPTION:
This is a post market study without interventions.The participants have been treated with CyPass-Stent implantation between 3 and 7 years ago to control the intraocular pressure . They will be invited for only one follow up visit to determine the present glaucoma status again, to determine the long term safety and effectiveness of the cypass stent procedure and to see whether addition therapy or surgical intervention is necessary.

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone a standalone cypass implantation at least 3 years ago
* signed inform consent

Exclusion Criteria:

* Patients with too much travel distance between study center and home
* Patients who cannot visit the studycenter due to health problems

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 130 Patient with at least one treated eye
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Hoeh, MD,FEBO, Principal Investigator — Department of Ophthalmology, Neubrandenburg, Germany
Locations (1):
- Dietrich-Bonhoeffer-Klinikum, Neubrandenburg, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: Yes
results will be published in ophthalmological journals
Time Frame: results are planned to published in December 2020
Access Criteria: Publication in ophthalmological journals provided and checked by Ahmed Medra

REFERENCES:
- [Background] Hoeh H, Vold SD, Ahmed IK, Anton A, Rau M, Singh K, Chang DF, Shingleton BJ, Ianchulev T. Initial Clinical Experience With the CyPass Micro-Stent: Safety and Surgical Outcomes of a Novel Supraciliary Microstent. J Glaucoma. 2016 Jan;25(1):106-12. doi: 10.1097/IJG.0000000000000134. PMID 25304276
- [Background] Garcia-Feijoo J, Rau M, Grisanti S, Grisanti S, Hoh H, Erb C, Guguchkova P, Ahmed I, Grabner G, Reitsamer H, Shaarawy T, Ianchulev T. Supraciliary Micro-stent Implantation for Open-Angle Glaucoma Failing Topical Therapy: 1-Year Results of a Multicenter Study. Am J Ophthalmol. 2015 Jun;159(6):1075-1081.e1. doi: 10.1016/j.ajo.2015.02.018. Epub 2015 Mar 3. PMID 25747677
- [Background] Grisanti S, Margolina E, Hoeh H, Rau M, Erb C, Kersten-Gomez I, Dick HB, Grisanti S. [Supraciliary microstent for open-angle glaucoma: clinical results of a prospective multicenter study]. Ophthalmologe. 2014 Jun;111(6):548-52. doi: 10.1007/s00347-013-2927-6. German. PMID 23958836
- [Background] Hoh H, Grisanti S, Grisanti S, Rau M, Ianchulev S. Two-year clinical experience with the CyPass micro-stent: safety and surgical outcomes of a novel supraciliary micro-stent. Klin Monbl Augenheilkd. 2014 Apr;231(4):377-81. doi: 10.1055/s-0034-1368214. Epub 2014 Apr 25. PMID 24771171

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standalone CyPass Implantation
Started | 230
Completed | 230
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: all patients that undergone a standalone Cypass-implantation
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 64
  >=65 years | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (12.095)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119
  Male | 111
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 230

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Achieve Target Intraocular Pressure Measured in mmHg
Description: The Measurement of the intraocular Pressure is a criterion for the Efficacy of CyPass Stent Procedure (success rate). The postoperative target pressure of 15 mmHg, 18 mmHg or 21 mmHg (depends on Glaucoma Status) has to be achieved.
Time Frame: up to 7 years
Population: only 75 study patients were able to visit the clinic and to undergone the 5 year examination, therefore we only could analyse the data of theses75 patients. The number of 230 Patients discribes all patients that fullfil the inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 75
Participants
  Target pressure achieved - without medication | 8
  Target pressure achieved - with medication | 45
  Target pressure not achieved | 22

2. Primary Outcome: Change of Intraocular Pressure in mmHg Preoperatively (at Screening) vs Postoperatively (at Final Examination)
Description: The Measurement of the intraocular Pressure change is a criterion for the Efficacy of CyPass Stent Procedure (success rate). The postoperative pressure after 5 to 7 years has to be compared with the preoperative intraocular pressure (in mmHg)
  The change was calculated only from two time points. (value at the final examination time point minus the value at the preoperative time point
Time Frame: up to 7 years
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 75
mmHg
  preoperative | 21.127 (7.831)
  postoperative | 16.553 (6.633)
  change | -4.697 (8.212)

3. Primary Outcome: Number of Additional Medication
Description: The number of additional Glaucoma medication is another criterion to determine the Efficacy of CyPass Stent Procedure (success rate). Up to 4 different active substance can be used to reduce the pressure. The more substances the patient uses postoperatively the lower is the success after implantation of the CyPass-Stent.
  The postoperative number of medications after 5 years has to be compared with the preoperative number
Time Frame: up to 7 years
Measure: Mean (Standard Deviation); unit: numbers of active substances
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 75
numbers of active substances
  preoperative | 1.813 (1.182)
  postoperative | 2.014 (1.053)
  change | 0.173 (1.201)

4. Primary Outcome: Number of Participants With Secondary Glaucoma Procedures
Description: To determine the efficacy of CyPass Stent procedure completely the number of secondary glaucoma interventions (surgery/ laser) has to be documented
Time Frame: up to 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 230
Participants | 83

5. Secondary Outcome: Number of Participants With Stability of Optic Nerve
Description: The Measurement of the optic nerve (HRT) in comparison to the baseline is needed to evaluate the glaucoma damage and to determine the Longterm success rate and the safety of the CyPass- Stent-Procedure.
  With papillary tomography you can see the changes in the optic nerve head concerning the permanent failures of retinal vessels , measure them very precisely and compare them with the previous findings.
Time Frame: up to 7 years
Population: for 7 eyes this examination was not done due to low compliance
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 68
Participants
  stable | 52
  not stable | 16

6. Secondary Outcome: Number of Participants With Stability of the Retinal Nerve Fiber Layer Thickness
Description: The comparison of the preoperative and postoperative Status of the Retinal Nerve Fiber Layer Thickness and retinal fundus thickness is another criterion to determine the absolute and relative success.
Time Frame: up to 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 75
Participants
  stable | 40
  worsening | 35

7. Secondary Outcome: Number of Participants With Stability of Visual Field
Description: The parameter of the Visual Field (Mean Deviation) will be measured to evaluate the Safety of the CyPass-Procedure. The visual Field shows the progression of glaucoma defects concerning failures in different parts for example in the center or in the periphery of the visual field.
Time Frame: up to 7 years
Population: The Overall Number of Participants Analyzed is not consistent with numbers provided in any of the rows in the Participant Flow module. The discrepancy is caused by insufficient cooperation (due to old age or poor general condition) of individual participants to carry out this examination to the end
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 73
Participants
  improvement | 11
  stable | 49
  progression | 13

8. Secondary Outcome: Number of Participants With Stability of Stent Position
Description: Determination of Stent Position in the angle will be performed to exclude moving of the Stent. The stent could change it's position forward into the anterior chamber or backwards in the suprachorioidal space
Time Frame: up to 7 years
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 68
Participants
  Stent is stable | 43
  Stent moves deeper | 12
  Stent emerges | 13

9. Secondary Outcome: Number of Participants With Stability of Stent Tissue Interaction
Description: Determination of iris tissue reaction to the stent will be performed. We document slight reaction without involving the opening, iris reaction with involving the opening and complete closure by tissue. The iris Tissue could overgrow the opening of the stent and therfore the function of the stent is disturbed or even failed.
Time Frame: up to 7 years
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 74
Participants
  stable | 24
  slight adhesions | 32
  severe adhesions | 18

10. Secondary Outcome: Number of Participants With Intra-and Postoperative Complications
Description: The number of intra-and postoperative complications are needed to evaluate the safety of the CyPass-procedure
Time Frame: up to 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 230
Participants
  resistance during implantation | 1
  heavy bleeding (intraoperative) | 6
  bad stent positioning | 5
  increase in pressure: early postoperative | 5
  increase in pressure | 25
  increase in pressure: glaucomatous attack | 17
  hyphema | 4
  hypotonia | 3
  early contact to the endothelium | 2
  age-related macula degeneration | 4
  gliosis | 2
  macula edema | 1
  keratitis | 1
  dry eyes symptoms | 5
  fibrin | 2
  stroke | 1
  uveitis | 1
  cataract progression | 15
  secondary cataract | 5
  lid tumor | 1
  pain during operation | 3
  recurrent neuritis | 1
  retroiridal cyst | 1
  total number of complications | 111
  total number of affected eyes | 105

11. Secondary Outcome: Number of Participants With Suprachoroidal Bleb
Description: The Determination of the suprachoroidal bleb is needed to evaluate the function of the stent and the efficacy of the procedure. The bigger the bleb, the lower the pressure and the better the efficacy of the stent
Time Frame: up to 7 years
Population: for 12 eyes this examination was not done due to low compliance
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone CyPass Implantation
Number analyzed (Participants) | 63
Participants
  none | 44
  small | 17
  big | 2

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Standalone CyPass Implantation: patients who have undergone a standalone cypass implantation without cataract surgery more than 3 years ago
  Glaucoma diagnostics: Heidelberg, Retinal Topography, Visual field, intraocular pressure, medication anamnesis, Retinal Nerve Fibre Layer Thickness, Pachymetry, Sonography, full ophthalmological determination
Arm/Group | Standalone CyPass Implantation
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 1/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standalone CyPass Implantation (N=75)
Allergic reaction (Eye disorders) | 1 (1) — itching, watery secretion, redning of the lids

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT03114059/Prot_SAP_000.pdf